CLINICAL TRIAL: NCT03922776
Title: Phenotypic Characterization Tumor-infiltrating Lymphocytes at Diagnosis and After Chemotherapy in Advanced High-grade Serous Ovarian Cancer in Blood, Ascites, Peritoneal Biopsy
Brief Title: Phenotypic Characterization Tumor-infiltrating Lymphocytes at Diagnosis and After Chemotherapy in Ovarian Cancer
Acronym: TILsOV-1805
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of recruiting period
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TILsOV-1805; Id RCB (Registry Identifier: 2018-A00771-54)
Record Dates: First submitted 2019-01-30; First posted 2019-04-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer Stage IIIC; Fallopian Tube Cancer Stage IIIC; Fallopian Tube Cancer Stage IV; Ovarian Cancer Stage IV
Keywords: Ovarian cancer; Tubal Cancer; Immunological profile; PBMc; TILs; Carcinomatosis; HGSOC
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood sample collection (Experimental): Participants will receive the following interventions because they are enrolled in the study: blood sample collection
  * at diagnosis, before chemotherapy (pre-CT)
  * after chemotherapy (post-ct)
  Intervention : Collection of two blood samples (5mL)
  * before chemotherapy (pre-CT), at diagnosis, up to 1 month after enrollment
  * and then, after chemotherapy (post-CT), up to 3 months after enrollment
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — Participants will receive the following interventions because they are enrolled in the study: blood sample collection
  * at diagnosis, before chemotherapy (pre-CT)
  * after chemotherapy (post-ct) Collection of two blood samples (5mL),
  * before chemotherapy (pre-CT), at diagnosis, up to 1 month after enrollment
  * and then, after chemotherapy (post-CT), up to 3 months after enrollment

SUMMARY:
This is a monocenter, interventional, non-randomized study among women patients with an ovarian or tubal cancer who will receive a surgery or adjuvant chemotherapy treatment, or a neo-adjuvant chemotherapy then surgery +/- adjuvant chemotherapy. The planned interventions are collection of biological samples at different times. The study will aim to describe the immunological profile at diagnosis in terms of phenotypic : PBMCs (peripheral blood, mononuclear cells) in peripheral blood, TILs (tumor-infiltrating lymphocytes) in ascites and in carcinomatosis.

DETAILED DESCRIPTION:
Participants will receive the following interventions because they are enrolled in the study: blood sample collection

* at diagnosis, before chemotherapy (pre-CT)
* after chemotherapy (post-ct)

Two additional blood samples will be collected in each patient : one at diagnosis and one at the end of chemotherapy.

The aim of this study is to describe the immunological profile at diagnosis in terms of phenotypic : PBMC in peripheral blood, TILs in ascites and in carcinomatosis, in patients treated for peritoneal carcinomatosis of ovarian or tubal origin. The treatment has to be a surgery and an adjuvant chemotherapy, or a neo-adjuvant chemotherapy followed by a surgery +/- adjuvant chemotherapy.

Other objectives of the study include:

* Evaluate the association between the immunological profile at diagnosis and the characteristics of the disease at diagnosis (histological type, extension)
* Evaluate the prognostic value of the immunological profile at diagnosis in terms of clinical response to neoadjuvant chemotherapy (for patients with interval surgery)
* Evaluate the polarization of the immune response induced by chemotherapy, describing the phenotypic changes in the different types of samples (blood, +/- ascites, +/- carcinomatosis) after chemotherapy in comparison with samples at diagnostic
* Evaluate the association between these immunological phenotypic changes and the clinical response to chemotherapy in patients receiving neoadjuvant chemotherapy
* Collect biological material for peritoneal carcinomatosis for subsequent biological analyzes

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Presenting a carcinomatosis with suspicion of ovarian cancer or tubal cancer, under a diagnostic laparoscopy
* Stage IIIC or initial pleural IV
* Planned treatment with surgery and adjuvant chemotherapy, or neo-adjuvant chemotherapy followed by surgery +/- adjuvant chemotherapy
* Having been informed and signed the informed consent of this study
* Affiliated with a social security scheme

Exclusion Criteria:

* Stage IV with visceral metastases (pulmonary, hepatic ...)
* Contraindication to surgery and / or chemotherapy
* Pregnant or lactating woman
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in a study of ovarian cancer
Enrollment: 36 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Counting of lymphocyte populations (pre-chemotherapy) | At diagnosis (during diagnostic laparoscopy, which is : before chemotherapy (pre-CT) and up to 1 month after enrollment)
  For each sample taken (blood / ascites / peritoneal carcinomatosis fragment), before chemotherapy, the lymphocyte populations will be counted by flow cytometry (CMF). For this, 4 panels of 32 markers will be used to identify 5 populations of lymphocytes: Thelper, B lymphocytes, TREG, TFH, TCD8, and immuno checkpoint
Counting of lymphocyte populations (post-chemotherapy) | At the end of chemotherapy (post-CT), up to 3 months
  For each sample taken (blood / ascites / peritoneal carcinomatosis fragment), at the end of chemotherapy, the lymphocyte populations will be counted by flow cytometry (CMF). For this, 4 panels of 32 markers will be used to identify 5 populations of lymphocytes: Thelper, B lymphocytes, TREG, TFH, TCD8, and immuno checkpoint

SECONDARY OUTCOMES:
Histological type on the initial biopsy | At diagnosis, before chemotherapy (pre-CT), up to 1 month after enrollment
  To check if there is an extension to the pleura (FIGO-IV) or not (FIGO-IIIC)
Clinical response to chemotherapy (post-chemotherapy) | At the end of chemotherapy, up to 3 months
  In patients receiving neo-adjuvant chemotherapy, clinical response to chemotherapy defined by a partial or complete radiological response (assessed on the thoraco-abdominopelvic CT scan), associated with a decrease in CA125 and a disappearance of ascites in case of ascites at inclusion
Histological response to chemotherapy (no residual disease on excised tissue) | At the surgery, an average of 6 weeks after inclusion
  Rate of patients with no residual disease on excised tissue regarding the assessment of histological response to chemotherapy
Progression-free survival | 6 months min to 14 months max
  Time between the diagnosis and the progression of the disease or the death of the patient, whatever the cause
Global survival | 6 months min to 14 months max
  Time between diagnosis and death, whatever the cause

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Hudry, MD, Principal Investigator — Département de cancérologie uro-digestive - Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bobisse S, Genolet R, Roberti A, Tanyi JL, Racle J, Stevenson BJ, Iseli C, Michel A, Le Bitoux MA, Guillaume P, Schmidt J, Bianchi V, Dangaj D, Fenwick C, Derre L, Xenarios I, Michielin O, Romero P, Monos DS, Zoete V, Gfeller D, Kandalaft LE, Coukos G, Harari A. Sensitive and frequent identification of high avidity neo-epitope specific CD8 + T cells in immunotherapy-naive ovarian cancer. Nat Commun. 2018 Mar 15;9(1):1092. doi: 10.1038/s41467-018-03301-0. PMID 29545564
- [Background] Zhang AW, McPherson A, Milne K, Kroeger DR, Hamilton PT, Miranda A, Funnell T, Little N, de Souza CPE, Laan S, LeDoux S, Cochrane DR, Lim JLP, Yang W, Roth A, Smith MA, Ho J, Tse K, Zeng T, Shlafman I, Mayo MR, Moore R, Failmezger H, Heindl A, Wang YK, Bashashati A, Grewal DS, Brown SD, Lai D, Wan ANC, Nielsen CB, Huebner C, Tessier-Cloutier B, Anglesio MS, Bouchard-Cote A, Yuan Y, Wasserman WW, Gilks CB, Karnezis AN, Aparicio S, McAlpine JN, Huntsman DG, Holt RA, Nelson BH, Shah SP. Interfaces of Malignant and Immunologic Clonal Dynamics in Ovarian Cancer. Cell. 2018 Jun 14;173(7):1755-1769.e22. doi: 10.1016/j.cell.2018.03.073. Epub 2018 May 10. PMID 29754820
- [Background] Mayor P, Starbuck K, Zsiros E. Adoptive cell transfer using autologous tumor infiltrating lymphocytes in gynecologic malignancies. Gynecol Oncol. 2018 Aug;150(2):361-369. doi: 10.1016/j.ygyno.2018.05.024. Epub 2018 May 24. PMID 29803316
- [Background] van Driel WJ, Koole SN, Sikorska K, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AGJ, Verwaal VJ, Kieffer JM, Van de Vijver KK, van Tinteren H, Aaronson NK, Sonke GS. Hyperthermic Intraperitoneal Chemotherapy in Ovarian Cancer. N Engl J Med. 2018 Jan 18;378(3):230-240. doi: 10.1056/NEJMoa1708618. PMID 29342393
- [Background] Odunsi K. Immunotherapy in ovarian cancer. Ann Oncol. 2017 Nov 1;28(suppl_8):viii1-viii7. doi: 10.1093/annonc/mdx444. PMID 29232467
- [Background] Tran E, Robbins PF, Rosenberg SA. 'Final common pathway' of human cancer immunotherapy: targeting random somatic mutations. Nat Immunol. 2017 Feb 15;18(3):255-262. doi: 10.1038/ni.3682. PMID 28198830
- [Background] Ovarian Tumor Tissue Analysis (OTTA) Consortium; Goode EL, Block MS, Kalli KR, Vierkant RA, Chen W, Fogarty ZC, Gentry-Maharaj A, Toloczko A, Hein A, Bouligny AL, Jensen A, Osorio A, Hartkopf A, Ryan A, Chudecka-Glaz A, Magliocco AM, Hartmann A, Jung AY, Gao B, Hernandez BY, Fridley BL, McCauley BM, Kennedy CJ, Wang C, Karpinskyj C, de Sousa CB, Tiezzi DG, Wachter DL, Herpel E, Taran FA, Modugno F, Nelson G, Lubinski J, Menkiszak J, Alsop J, Lester J, Garcia-Donas J, Nation J, Hung J, Palacios J, Rothstein JH, Kelley JL, de Andrade JM, Robles-Diaz L, Intermaggio MP, Widschwendter M, Beckmann MW, Ruebner M, Jimenez-Linan M, Singh N, Oszurek O, Harnett PR, Rambau PF, Sinn P, Wagner P, Ghatage P, Sharma R, Edwards RP, Ness RB, Orsulic S, Brucker SY, Johnatty SE, Longacre TA, Ursula E, McGuire V, Sieh W, Natanzon Y, Li Z, Whittemore AS, Anna A, Staebler A, Karlan BY, Gilks B, Bowtell DD, Hogdall E, Candido dos Reis FJ, Steed H, Campbell IG, Gronwald J, Benitez J, Koziak JM, Chang-Claude J, Moysich KB, Kelemen LE, Cook LS, Goodman MT, Garcia MJ, Fasching PA, Kommoss S, Deen S, Kjaer SK, Menon U, Brenton JD, Pharoah PDP, Chenevix-Trench G, Huntsman DG, Winham SJ, Kobel M, Ramus SJ. Dose-Response Association of CD8+ Tumor-Infiltrating Lymphocytes and Survival Time in High-Grade Serous Ovarian Cancer. JAMA Oncol. 2017 Dec 1;3(12):e173290. doi: 10.1001/jamaoncol.2017.3290. PMID 29049607
- [Background] Delcourt V, Franck J, Leblanc E, Narducci F, Robin YM, Gimeno JP, Quanico J, Wisztorski M, Kobeissy F, Jacques JF, Roucou X, Salzet M, Fournier I. Combined Mass Spectrometry Imaging and Top-down Microproteomics Reveals Evidence of a Hidden Proteome in Ovarian Cancer. EBioMedicine. 2017 Jul;21:55-64. doi: 10.1016/j.ebiom.2017.06.001. Epub 2017 Jun 3. PMID 28629911
- [Background] Murakami R, Matsumura N, Mandai M, Yoshihara K, Tanabe H, Nakai H, Yamanoi K, Abiko K, Yoshioka Y, Hamanishi J, Yamaguchi K, Baba T, Koshiyama M, Enomoto T, Okamoto A, Murphy SK, Mori S, Mikami Y, Minamiguchi S, Konishi I. Establishment of a Novel Histopathological Classification of High-Grade Serous Ovarian Carcinoma Correlated with Prognostically Distinct Gene Expression Subtypes. Am J Pathol. 2016 May;186(5):1103-13. doi: 10.1016/j.ajpath.2015.12.029. Epub 2016 Mar 15. PMID 26993207
- [Background] Blank CU, Haanen JB, Ribas A, Schumacher TN. CANCER IMMUNOLOGY. The "cancer immunogram". Science. 2016 May 6;352(6286):658-60. doi: 10.1126/science.aaf2834. No abstract available. PMID 27151852
- [Background] Santoiemma PP, Powell DJ Jr. Tumor infiltrating lymphocytes in ovarian cancer. Cancer Biol Ther. 2015;16(6):807-20. doi: 10.1080/15384047.2015.1040960. Epub 2015 Apr 20. PMID 25894333
- [Background] Hiraoka N, Ino Y, Yamazaki-Itoh R, Kanai Y, Kosuge T, Shimada K. Intratumoral tertiary lymphoid organ is a favourable prognosticator in patients with pancreatic cancer. Br J Cancer. 2015 May 26;112(11):1782-90. doi: 10.1038/bjc.2015.145. Epub 2015 May 5. PMID 25942397
- [Background] Salgado R, Denkert C, Demaria S, Sirtaine N, Klauschen F, Pruneri G, Wienert S, Van den Eynden G, Baehner FL, Penault-Llorca F, Perez EA, Thompson EA, Symmans WF, Richardson AL, Brock J, Criscitiello C, Bailey H, Ignatiadis M, Floris G, Sparano J, Kos Z, Nielsen T, Rimm DL, Allison KH, Reis-Filho JS, Loibl S, Sotiriou C, Viale G, Badve S, Adams S, Willard-Gallo K, Loi S; International TILs Working Group 2014. The evaluation of tumor-infiltrating lymphocytes (TILs) in breast cancer: recommendations by an International TILs Working Group 2014. Ann Oncol. 2015 Feb;26(2):259-71. doi: 10.1093/annonc/mdu450. Epub 2014 Sep 11. PMID 25214542
- [Background] Galluzzi L, Vacchelli E, Bravo-San Pedro JM, Buque A, Senovilla L, Baracco EE, Bloy N, Castoldi F, Abastado JP, Agostinis P, Apte RN, Aranda F, Ayyoub M, Beckhove P, Blay JY, Bracci L, Caignard A, Castelli C, Cavallo F, Celis E, Cerundolo V, Clayton A, Colombo MP, Coussens L, Dhodapkar MV, Eggermont AM, Fearon DT, Fridman WH, Fucikova J, Gabrilovich DI, Galon J, Garg A, Ghiringhelli F, Giaccone G, Gilboa E, Gnjatic S, Hoos A, Hosmalin A, Jager D, Kalinski P, Karre K, Kepp O, Kiessling R, Kirkwood JM, Klein E, Knuth A, Lewis CE, Liblau R, Lotze MT, Lugli E, Mach JP, Mattei F, Mavilio D, Melero I, Melief CJ, Mittendorf EA, Moretta L, Odunsi A, Okada H, Palucka AK, Peter ME, Pienta KJ, Porgador A, Prendergast GC, Rabinovich GA, Restifo NP, Rizvi N, Sautes-Fridman C, Schreiber H, Seliger B, Shiku H, Silva-Santos B, Smyth MJ, Speiser DE, Spisek R, Srivastava PK, Talmadge JE, Tartour E, Van Der Burg SH, Van Den Eynde BJ, Vile R, Wagner H, Weber JS, Whiteside TL, Wolchok JD, Zitvogel L, Zou W, Kroemer G. Classification of current anticancer immunotherapies. Oncotarget. 2014 Dec 30;5(24):12472-508. doi: 10.18632/oncotarget.2998. PMID 25537519
- [Background] Tangye SG, Ma CS, Brink R, Deenick EK. The good, the bad and the ugly - TFH cells in human health and disease. Nat Rev Immunol. 2013 Jun;13(6):412-26. doi: 10.1038/nri3447. Epub 2013 May 17. PMID 23681096
- [Background] Bachmayr-Heyda A, Aust S, Heinze G, Polterauer S, Grimm C, Braicu EI, Sehouli J, Lambrechts S, Vergote I, Mahner S, Pils D, Schuster E, Thalhammer T, Horvat R, Denkert C, Zeillinger R, Castillo-Tong DC. Prognostic impact of tumor infiltrating CD8+ T cells in association with cell proliferation in ovarian cancer patients--a study of the OVCAD consortium. BMC Cancer. 2013 Sep 17;13:422. doi: 10.1186/1471-2407-13-422. PMID 24044611
- [Background] Aghajanian C, Blank SV, Goff BA, Judson PL, Teneriello MG, Husain A, Sovak MA, Yi J, Nycum LR. OCEANS: a randomized, double-blind, placebo-controlled phase III trial of chemotherapy with or without bevacizumab in patients with platinum-sensitive recurrent epithelial ovarian, primary peritoneal, or fallopian tube cancer. J Clin Oncol. 2012 Jun 10;30(17):2039-45. doi: 10.1200/JCO.2012.42.0505. Epub 2012 Apr 23. PMID 22529265
- [Background] Hwang WT, Adams SF, Tahirovic E, Hagemann IS, Coukos G. Prognostic significance of tumor-infiltrating T cells in ovarian cancer: a meta-analysis. Gynecol Oncol. 2012 Feb;124(2):192-8. doi: 10.1016/j.ygyno.2011.09.039. Epub 2011 Oct 29. PMID 22040834
- [Background] Burger RA, Brady MF, Bookman MA, Fleming GF, Monk BJ, Huang H, Mannel RS, Homesley HD, Fowler J, Greer BE, Boente M, Birrer MJ, Liang SX; Gynecologic Oncology Group. Incorporation of bevacizumab in the primary treatment of ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2473-83. doi: 10.1056/NEJMoa1104390. PMID 22204724
- [Background] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Background] Sato E, Olson SH, Ahn J, Bundy B, Nishikawa H, Qian F, Jungbluth AA, Frosina D, Gnjatic S, Ambrosone C, Kepner J, Odunsi T, Ritter G, Lele S, Chen YT, Ohtani H, Old LJ, Odunsi K. Intraepithelial CD8+ tumor-infiltrating lymphocytes and a high CD8+/regulatory T cell ratio are associated with favorable prognosis in ovarian cancer. Proc Natl Acad Sci U S A. 2005 Dec 20;102(51):18538-43. doi: 10.1073/pnas.0509182102. Epub 2005 Dec 12. PMID 16344461
- [Background] Curiel TJ, Coukos G, Zou L, Alvarez X, Cheng P, Mottram P, Evdemon-Hogan M, Conejo-Garcia JR, Zhang L, Burow M, Zhu Y, Wei S, Kryczek I, Daniel B, Gordon A, Myers L, Lackner A, Disis ML, Knutson KL, Chen L, Zou W. Specific recruitment of regulatory T cells in ovarian carcinoma fosters immune privilege and predicts reduced survival. Nat Med. 2004 Sep;10(9):942-9. doi: 10.1038/nm1093. Epub 2004 Aug 22. PMID 15322536
- [Background] Zhang L, Conejo-Garcia JR, Katsaros D, Gimotty PA, Massobrio M, Regnani G, Makrigiannakis A, Gray H, Schlienger K, Liebman MN, Rubin SC, Coukos G. Intratumoral T cells, recurrence, and survival in epithelial ovarian cancer. N Engl J Med. 2003 Jan 16;348(3):203-13. doi: 10.1056/NEJMoa020177. PMID 12529460
- [Background] Dunn GP, Bruce AT, Ikeda H, Old LJ, Schreiber RD. Cancer immunoediting: from immunosurveillance to tumor escape. Nat Immunol. 2002 Nov;3(11):991-8. doi: 10.1038/ni1102-991. PMID 12407406